CLINICAL TRIAL: NCT01708668
Title: The Effects of Intermittent Epidural Bolus Versus Continuous Epidural Infusion on Fever for Labor Analgesia in Primiparous Women
Brief Title: The Effects of Intermittent Epidural Bolus on Fever During Labor Analgesia
Acronym: EIEBFLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ShanWu Feng, M.D. (Other)
Responsible Party: Sponsor-Investigator, ShanWu Feng, M.D., Department of Anesthesiology, Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China, 210004, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NJMCHH-2012-A010; 08NMUM063 (Other Grant/Funding Number: Nanjing Medical University); YKK08119 (Other Grant/Funding Number: Nanjing Department of Health); YKK11058 (Other Grant/Funding Number: Nanjing Department of Health)
Record Dates: First submitted 2012-10-07; First posted 2012-10-17 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Labor Pain; Pain; Neurologic Manifestations; Signs and Symptoms; Pathological Conditions, Signs and Symptoms
Keywords: Fever; Patient controlled epidural analgesia; Labor analgesia; Epidural analgesia; Combined spinal-epidural analgesia
MeSH Terms: conditions — Labor Pain; Pain; Neurologic Manifestations; Signs and Symptoms; Pathological Conditions, Signs and Symptoms; Fever | interventions — Analgesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1 (Active Comparator): Epidural analgesia (EA) with continuous epidural infusion(CEI)
  Interventions: Procedure: Epidural analgesia; Procedure: Continuous epidural infusion
- 2 (Active Comparator): Combined spinal-epidural analgesia (CSEA) with continuous epidural infusion(CEI)
  Interventions: Procedure: Combined spinal-epidural analgesia; Procedure: Continuous epidural infusion
- 3 (Active Comparator): Epidural analgesia (EA) with intermittent epidural bolus (IEB, 2.5 mL bolused every 15 minutes)
  Interventions: Procedure: Epidural analgesia; Procedure: Intermittent epidural bolus
- 4 (Active Comparator): Epidural analgesia (EA) with intermittent epidural bolus (IEB, 5ml bolused every 30 minutes)
  Interventions: Procedure: Epidural analgesia; Procedure: Intermittent epidural bolus
- 5 (Active Comparator): Epidural analgesia (EA) with intermittent epidural bolus (IEB, 10ml bolused every 60 minutes)
  Interventions: Procedure: Epidural analgesia; Procedure: Intermittent epidural bolus
- 6 (Active Comparator): Combined spinal-epidural analgesia (CSEA) with intermittent epidural bolus (IEB, 2.5 mL bolused every 15 minutes)
  Interventions: Procedure: Combined spinal-epidural analgesia; Procedure: Intermittent epidural bolus
- 7 (Active Comparator): Combined spinal-epidural analgesia (CSEA) with intermittent epidural bolus (IEB, 5ml bolused every 30 minutes)
  Interventions: Procedure: Combined spinal-epidural analgesia; Procedure: Intermittent epidural bolus
- 8 (Active Comparator): Combined spinal-epidural analgesia (CSEA) with intermittent epidural bolus (IEB, 10ml bolused every 60 minutes)
  Interventions: Procedure: Combined spinal-epidural analgesia; Procedure: Intermittent epidural bolus

INTERVENTIONS:
Procedure: Epidural analgesia
  Arms: 1; 3; 4; 5
Procedure: Combined spinal-epidural analgesia
  Arms: 2; 6; 7; 8
Procedure: Continuous epidural infusion
  Arms: 1; 2
Procedure: Intermittent epidural bolus
  Arms: 3; 4; 5; 6; 7; 8

SUMMARY:
Epidural analgesia is associated with maternal intra-partum fever during labor. Intermittent epidural injections appear to reduce the incidence of maternal intra-partum fever compared to continuous epidural infusion during labor analgesia. However, the optimal combination of bolus volume and administrating interval has not yet been compared. The purpose of this prospective, randomized, double-blind trial was to determine how intermittent epidural bolus reduced the incidence of maternal intra-partum fever compared with continuous epidural infusion during labor.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Required labor analgesia
* Chinese
* Spontaneous labor

Exclusion Criteria:

* Contraindications for epidural analgesia
* Allergic to opioids and/or local anesthetics
* Failed to performing epidural catheterization
* Organic dysfunction
* Those who were not willing to or could not finish the whole study at any time
* Using or used in the past 14 days of the monoamine oxidase inhibitors
* Alcohol addictive or narcotic dependent patients
* Subjects with a nonvertex presentation or scheduled induction of labor
* Twin gestation and breech presentation

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12000 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-07 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Maternal oral and tympanic temperature | At time of initiation of analgesia and hourly thereafter until 4 hours postpartum (approximately 12 hours)

SECONDARY OUTCOMES:
Maternal serum Interleukin-1β | At time of placental delivery and 3, 6 and 12 hours later
Cord serum Interleukin-1β | At time of placental delivery
Maternal serum Interleukin-6 | At time of placental delivery and 3, 6 and 12 hours later
Cord serum Interleukin-6 | At time of placental delivery
Maternal serum Interleukin-10 | At time of placental delivery and 3, 6 and 12 hours later
Cord serum Interleukin-10 | At time of placental delivery
Maternal serum tumor necrosis factor-α | At time of placental delivery and 3, 6 and 12 hours later
Cord serum tumor necrosis factor-α | At time of placental delivery
Regression and correlation analyses between maternal and cord serum cytokines | At twelve hours postpartum
Placental routine pathologic examination | At time of placental delivery
Maternal and cord blood gase analysis | At time of placental delivery
Maternal modified Bromage scale and visual analogue scale | At time of initiation of analgesia and hourly thereafter until 2 hours postpartum (approximately 10 hours)
Rescue boluses, n of rescue boluses, and the consumption of the ropivacaine/sufentanil mixture | At two hours postpartum
Rates of cesarean delivery and instrument-assisted delivery | At time of placental delivery
Indications of cesarean delivery | Initiation of analgesia to placental delivery (approximately 8 hours)
Duration of analgesia | Initiation of analgesia to 2 h postpartum (approximately 10 hours)
Durations of labor stages | From the beginning of regular contraction of uterus to the end of the labor (approximately 12 hours)
Maternal satisfaction with analgesia | At two hours postpartum
Use of oxytocin after analgesia | At twenty-four hours postpartum
Low back pain at 3 months after vaginal delivery | At the third month after vaginal delivery
Breastfeeding success at 6 weeks after vaginal delivery | At the sixth week after successful delivery
Neonatal Apgar scale | At the first and fifth minutes after baby was born
Incidence of maternal side effects | Initiation of analgesia to 2 hour postpartum (approximately 10 hours)
Neonatal Neurologic and Adaptive Capacity Score | At 30 min, 2 h, and 24 h after baby was born
Maximal oxytocin dose | At twenty-four hours postpartum
Neonatal sepsis evaluation | At 30 min after baby was born
Neonatal antibiotic treatment | One week after baby was born
Maternal heart rate, respiratory rate, and blood pressure | At time of initiation of analgesia and hourly thereafter until 4 hours postpartum (approximately 12 hours)
Highest thoracic sensory level to alcohol | At three hours after initiation of analgesia
Uterine contraction | At time of initiation of analgesia and hourly thereafter until 4 hours postpartum (approximately 12 hours)
Neonatal rectal temperature | At delivery, 30 min after delivery, and 1 h after delivery
Fetal heart rate | From initiation of analgesia to delivery (approximately 8 hours)
Maternal group B streptococcus (GBS) colonization | At time of initiation of analgesia
Number of vaginal examinations, duration from rupture of the membranes to delivery, mode of membranes ruptured | From initiation of analgesia to delivery (approximately 8 hours)
Neonatal weight | At delivery
Uterine artery, umbilical artery and vein, fetus middle cerebral artery by ultrasound | At time of initiation of analgesia and hourly thereafter until delivery (approximately 8 hours)
Maternal serum epinephrine, norepinephrine, insulin, glucagon, corticotropin releasing hormone, adrenocorticotropic hormone, cortisol, blood glucose, oxytocin, prostaglandin E2 and prostaglandin F2 alpha | At time of initiation of analgesia and hourly thereafter until 4 hours postpartum (approximately 12 hours)
Maternal postpartum depression | At time of delivery and daily thereafter until 1 year postpartum (approximately 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Shanwu Feng, M.D., Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu, China